CLINICAL TRIAL: NCT00838877
Title: Open Label Positron Emission Tomography Study With [18F]AZD4694 and [11C]AZD2184, Candidate Radioligands for AB Amyloid, to Determine and Compare in Vivo Brain Uptake and Distribution in Healthy Volunteers and Patients With Alzheimer's Disease
Brief Title: Positron Emission Tomography (PET) Study With [18F]AZD4694 and [11C]AZD2184, Candidate PET Ligands for Aβ Amyloid
Acronym: PET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Björn Paulsson, MD, Medical Science Director, AD & Cognition, AstraZeneca R&D Södertälje, Sweden
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D2750C00001; 2008-006747-39
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2009-10-23 (Estimated); Status verified 2009-10

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; PET; Phase 1; Positron Emission Tomography
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: radioligand [18F]AZD4694; Drug: radioligand [11C]AZD2184

INTERVENTIONS:
Drug: radioligand [18F]AZD4694 — single dose of iv. admin. 1-2 times per subject
Drug: radioligand [11C]AZD2184 — single dose of iv admin. 1 time per subject

SUMMARY:
The study is carried out in order to investigate if [18F]AZD4694, compared to [11C]AZD2184, is a suitable PET ligand for in vivo imaging of Aβ amyloid depositions in the human brain. In the study the two PET ligands will be examined in both healthy volunteers and patients with Alzheimer's Disease. A whole body dosimetry scanning will be performed in 6 healthy volunteers to obtain human data to estimate a safe dose.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's Disease patients - 50-85 years, mild to moderate AD: MMSE ≥16 and ≤ 26, clinical progression of AD over 12 months.
* Healthy volunteers: - 50-75 years
* BMI 18 and 30 m2/kg
* Clinically normal physical findings including supine blood pressure and pulse rate.

Exclusion Criteria:

* Alzheimer's Disease patients - Clinically significant illness the 2 weeks prior to the administration of the PET ligand
* Significant cerebrovascular disease or depression, central nervous system infarct or infection or lesions
* Administration of any investigational product within 3 months prior to study and/or PET measurements for scientific purposes within the last 12 months.
* Healthy volunteers - clinically significant illness within 2 weeks before administration of PET ligand, history of psychiatric or somatic disease/condition that may interfere, first degree relative with dementia. Obvious deterioration of memory functions.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2009-01; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Positron emission tomography using the radioligand [18F]AZD4694 and/or [11C]AZD2184 | Radioligand [18F]AZD4694: 1-2 PET examinations for AD patients and 1 PET examination for healthy volunteers. Whole body dosimetri for some healthy volunteers. - Radioligand [11C]AZD2184: 1 PET for AD patients respective healthy volunteers.

SECONDARY OUTCOMES:
To assess safety and tolerability of [18F]AZD4694 and the study procedures, by assessment of adverse events, vital signs, and laboratory variables. | 3-4 visits with tests for AD patients respective healthy volunteers. All tests are not done at every visit.

CONTACTS AND LOCATIONS:
Overall Officials: Maria E Jönhagen, Principal Investigator — Geriatric Clinic, Karolinska University Hospital, Huddinge, Sweden; Ingemar Bylesjö, Principal Investigator — AstraZeneca Clinical Pharmacology Unit, Stockholm; Per Julin, Study Chair — AstraZeneca R&D, Södertälje, Sweden
Locations (2):
- Sweden (2):
  - Research Site, Huddinge
  - Research Site, Stockholm